CLINICAL TRIAL: NCT00145925
Title: ADVANCE - Action in Diabetes and Vascular Disease: Preterax and Diamicron - MR Controlled Evaluation
Brief Title: Blood Pressure and Glucose Lowering for the Prevention of Vascular Disease in High Risk Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: Institut de Recherches Internationales Servier (Other); University of Sydney (Other); National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: ADVANCE
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2008-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Blood Pressure; Stroke; MI
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Stroke | interventions — indapamide, perindopril drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blood pressure (Placebo Comparator): Perindopril indapamide vs placebo
  Interventions: Drug: Perindopril-indapamide
- Glucose control (Other): Standard versus intensive glucose control
  Interventions: Drug: Gliclazide MR-based glucose lowering

INTERVENTIONS:
Drug: Perindopril-indapamide
  Arms: Blood pressure
Drug: Gliclazide MR-based glucose lowering
  Arms: Glucose control

SUMMARY:
The purpose of this study is to provide information on the risks and benefits of routine blood pressure lowering (regardless of blood pressure level), and intensive lowering of blood glucose levels, in patients with Type 2 diabetes at high risk of cardiovascular events. The major outcomes of the study will be cardiovascular events (heart attack, stroke or dying as a result of cardiovascular disease), as well as new or worsening diabetic eye and kidney disease.

DETAILED DESCRIPTION:
Patients with type 2 diabetes are at increased risks of macrovascular and microvascular disease, both of which are reduced by control of raised blood pressure in hypertensive individuals. Intensive glycaemic control has also been shown to reduce microvascular disease, but the effects on macrovascular disease remain uncertain. This study will examine the hypotheses that blood pressure lowering (with an ACE inhibitor-diuretic combination) and intensive glycaemic control (with a sulphonylurea-based regimen) in high-risk individuals with type 2 diabetes (including hypertensive and non-hypertensive subjects) reduces the incidence of both macrovascular and microvascular disease.

The study is a 2 x 2 factorial randomised controlled trial that includes 11,140 adults with type 2 diabetes at elevated risk of vascular disease. Following 6 weeks on open label perindopril-indapamide combination, eligible individuals were randomised to continued perindopril-indapamide or matching placebo, and to an intensive gliclazide MR-based glucose control regimen (aiming for HbA1c of 6.5% or lower) or usual guidelines-based therapy. Primary outcomes are, first, the composite of non-fatal stroke, non-fatal myocardial infarction or cardiovascular death and, second, the composite of new or worsening nephropathy or diabetic eye disease. These primary outcomes will be analysed jointly and separately. The average duration of treatment and follow-up is 5.5 to 6 years. The study is being conducted in 214 centres in Australasia, Asia, Europe and North America.

ADVANCE is designed to provide reliable evidence about the balance of benefits and risks conferred by blood pressure lowering therapy and intensive glucose control therapy in high-risk diabetic patients, irrespective of initial blood pressure or glucose levels.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of type 2 diabetes mellitus first made at age 30 years or older
2. Age 55 years or older at entry
3. Ability to provide informed consent
4. A substantially elevated risk of cardiovascular disease, indicated by:

   * A history of major macrovascular disease defined as any one of: stroke, myocardial infarction, hospital admission for transient ischaemic attack, hospital admission for unstable angina, coronary artery bypass graft, percutaneous transluminal coronary angioplasty (with or without stenting), peripheral revascularisation (angioplasty or surgery) or amputation secondary to vascular disease or
   * A history of major microvascular disease defined as any one of nephropathy (albumin:creatinine ratio >300ug/mg), retinal photocoagulation therapy, proliferative retinopathy (new blood vessels on the disc or elsewhere, vitreous haemorrhage, pre-retinal haemorrhage, or fibrous proliferations on the disc or elsewhere), macular oedema (retinal thickening within one disc diameter of the macular centre) or blindness in either eye (corrected visual acuity 6/60 or worse, persisting for three months or more) not known to be due to non-diabetic causes or
   * A first diagnosis of type 2 diabetes made 10 or more years prior to entry or
   * Another major risk factor for vascular disease defined as any one of: current daily cigarette smoking, total cholesterol greater than 6.0 mmol/l (with or without cholesterol lowering treatment), HDL cholesterol <1.0 mmol/l, microalbuminuria (albumin:creatinine ratio 30-300ug/mg) or
   * Age 65 years or over

Exclusion Criteria:

1. A definite contraindication to treatment with an ACE inhibitor or a thiazide-like diuretic
2. A specific indication for treatment with an ACE inhibitor other than perindopril 2-4 mg daily (see also section 5.2.3) or a thiazide-like diuretic
3. A definite and specific indication for treatment with gliclazide or a haemoglobin A1c control target of 6.5% or less
4. A definite contra-indication to treatment with gliclazide or a haemoglobin A1c control target of 6.5% or less
5. A definite indication for long-term full-dose or bed-time insulin therapy
6. Participation in a trial within the month prior to the Registration Visit or current participation in another trial

Other potential reasons for ineligibility include:

* High probability of non-adherence to study treatment or follow-up
* Current clinical instability (e.g. a major cerebral or coronary event or sight-threatening retinopathy or macular oedema within the previous few weeks)
* Life threatening non-vascular disease other than diabetes and its complications
* Moderate or severe dementia
* Major disability that is likely to prevent regular attendance at study clinics

Final decisions about eligibility were made at the discretion of the study investigator and the potential study participant, in the light of any requirements or guidance from local ethics committees and other regulatory bodies.

Ages: 55 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11140 (Actual)
Dates: Start 2001-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Composite of non-fatal stroke, non-fatal myocardial infarction or death from any cardiovascular cause | July 2001 - December 2007
Composite of new or substantially worsening nephropathy or microvascular eye disease. | July 2001 - December 2007

SECONDARY OUTCOMES:
Includes cerebrovascular disease, coronary heart disease, heart failure, peripheral vascular disease, cardiovascular and all-cause mortality, microalbuminuria, visual deterioration, new or worsening nephropathy, cognitive function, and dementia. | July 2001 - December 2007

CONTACTS AND LOCATIONS:
Overall Officials: John Chalmers, MB BS PhD, Principal Investigator — The George Institute; Stephen W MacMahon, BSc PhD MPH, Principal Investigator — The George Institute
Locations (5):
- The University of Melbourne, Melbourne, Victoria, Australia
- University of Montreal, Montreal, Quebec, Canada
- Cardiovascular Institute & Fu Wai Hospital, Beijing, Beijing Municipality, China
- The Julius Center for Health Sciences and Primary Care, Utrecht, Utrecht, Netherlands
- Imperial College School of Medicine, London, United Kingdom

REFERENCES:
- [Background] Rationale and design of the ADVANCE study: a randomised trial of blood pressure lowering and intensive glucose control in high-risk individuals with type 2 diabetes mellitus. Action in Diabetes and Vascular Disease: PreterAx and DiamicroN Modified-Release Controlled Evaluation. J Hypertens Suppl. 2001 Nov;19(4):S21-8. PMID 11848259
- [Background] ADVANCE Collaborative Group. ADVANCE--Action in Diabetes and Vascular Disease: patient recruitment and characteristics of the study population at baseline. Diabet Med. 2005 Jul;22(7):882-8. doi: 10.1111/j.1464-5491.2005.01596.x. PMID 15975103
- [Background] ADVANCE Management Committee. Study rationale and design of ADVANCE: action in diabetes and vascular disease--preterax and diamicron MR controlled evaluation. Diabetologia. 2001 Sep;44(9):1118-20. doi: 10.1007/s001250100612. PMID 11596665
- [Derived] Harris K, Gong J, MacMahon S, Xu Y, Shajahan S, Harrap S, Poulter N, Marre M, Hamet P, Mancia G, Anderson C, Woodward M, Chalmers J. Effect of randomised blood pressure lowering treatment and intensive glucose control on dementia and cognitive decline according to baseline cognitive function and other subpopulations of individuals with type 2 diabetes: Results from the ADVANCE trial. Cereb Circ Cogn Behav. 2024 Dec 5;8:100372. doi: 10.1016/j.cccb.2024.100372. eCollection 2025. PMID 39758508
- [Derived] Wang N, Harris K, Woodward M, Harrap S, Mancia G, Poulter N, Chalmers J, Rodgers A; PROGRESS and ADVANCE collaborators. Clinical Utility of Short-Term Blood Pressure Measures to Inform Long-Term Blood Pressure Management. Hypertension. 2023 Mar;80(3):608-617. doi: 10.1161/HYPERTENSIONAHA.122.20458. Epub 2022 Dec 5. PMID 36468403
- [Derived] Ohkuma T, Harris K, Cooper M, Grobbee DE, Hamet P, Harrap S, Mancia G, Marre M, Patel A, Rodgers A, Williams B, Woodward M, Chalmers J; ADVANCE Collaborative Group. Short-Term Changes in Serum Potassium and the Risk of Subsequent Vascular Events and Mortality: Results from a Randomized Controlled Trial of ACE Inhibitors. Clin J Am Soc Nephrol. 2022 Aug;17(8):1139-1149. doi: 10.2215/CJN.00180122. Epub 2022 Jul 27. PMID 35896277
- [Derived] Juraschek SP, Wang D, McEvoy JW, Harrap S, Harris K, Mancia G, Marre M, Neal B, Patel A, Poulter NR, Williams B, Chalmers J, Woodward M, Selvin E. Effects of glucose and blood pressure reduction on subclinical cardiac damage: Results from ADVANCE. Int J Cardiol. 2022 Jul 1;358:103-109. doi: 10.1016/j.ijcard.2022.04.044. Epub 2022 Apr 18. PMID 35439582
- [Derived] Harris K, Muntner P, Woodward M, Jun M, Oshima M, Gong J, Harrap S, Menard J, Chalmers J. Clinical outcomes by atherosclerotic cardiovascular disease risk score and blood pressure level in high risk individuals with type 2 diabetes. J Hum Hypertens. 2023 Mar;37(3):181-188. doi: 10.1038/s41371-022-00661-5. Epub 2022 Feb 19. PMID 35184142
- [Derived] Nguyen TN, Harris K, Woodward M, Chalmers J, Cooper M, Hamet P, Harrap S, Heller S, MacMahon S, Mancia G, Marre M, Poulter N, Rogers A, Williams B, Zoungas S, Chow CK, Lindley RI. The Impact of Frailty on the Effectiveness and Safety of Intensive Glucose Control and Blood Pressure-Lowering Therapy for People With Type 2 Diabetes: Results From the ADVANCE Trial. Diabetes Care. 2021 Jul;44(7):1622-1629. doi: 10.2337/dc20-2664. Epub 2021 May 25. PMID 34035077
- [Derived] Wang N, Harris K, Chalmers J, Harrap S, Mancia G, Marre M, Poulter N, Tzourio C, Williams B, Zoungas S, Woodward M, Rodgers A. Combination blood pressure lowering in the presence or absence of background statin and aspirin therapy: a combined analysis of PROGRESS and ADVANCE Trials. J Hypertens. 2021 Aug 1;39(8):1689-1696. doi: 10.1097/HJH.0000000000002862. PMID 33883461
- [Derived] Gong J, Harris K, Hackett M, Peters SAE, Brodaty H, Cooper M, Hamet P, Harrap S, Mancia G, MacMahon S, Chalmers J, Woodward M. Sex differences in risk factors for cognitive decline and dementia, including death as a competing risk, in individuals with diabetes: Results from the ADVANCE trial. Diabetes Obes Metab. 2021 Aug;23(8):1775-1785. doi: 10.1111/dom.14391. Epub 2021 May 4. PMID 33783955
- [Derived] Tham YK, Jayawardana KS, Alshehry ZH, Giles C, Huynh K, Smith AAT, Ooi JYY, Zoungas S, Hillis GS, Chalmers J, Meikle PJ, McMullen JR. Novel Lipid Species for Detecting and Predicting Atrial Fibrillation in Patients With Type 2 Diabetes. Diabetes. 2021 Jan;70(1):255-261. doi: 10.2337/db20-0653. Epub 2020 Oct 28. PMID 33115826
- [Derived] Harris K, Oshima M, Sattar N, Wurtz P, Jun M, Welsh P, Hamet P, Harrap S, Poulter N, Chalmers J, Woodward M. Plasma fatty acids and the risk of vascular disease and mortality outcomes in individuals with type 2 diabetes: results from the ADVANCE study. Diabetologia. 2020 Aug;63(8):1637-1647. doi: 10.1007/s00125-020-05162-z. Epub 2020 May 8. PMID 32385604
- [Derived] Tian J, Ohkuma T, Cooper M, Harrap S, Mancia G, Poulter N, Wang JG, Zoungas S, Woodward M, Chalmers J. Effects of Intensive Glycemic Control on Clinical Outcomes Among Patients With Type 2 Diabetes With Different Levels of Cardiovascular Risk and Hemoglobin A1c in the ADVANCE Trial. Diabetes Care. 2020 Jun;43(6):1293-1299. doi: 10.2337/dc19-1817. Epub 2020 Mar 19. PMID 32193249
- [Derived] Oshima M, Jun M, Ohkuma T, Toyama T, Wada T, Cooper ME, Hadjadj S, Hamet P, Harrap S, Mancia G, Marre M, Williams B, Chalmers J, Woodward M, Perkovic V; ADVANCE Collaborative Group. The relationship between eGFR slope and subsequent risk of vascular outcomes and all-cause mortality in type 2 diabetes: the ADVANCE-ON study. Diabetologia. 2019 Nov;62(11):1988-1997. doi: 10.1007/s00125-019-4948-4. Epub 2019 Jul 13. PMID 31302707
- [Derived] Ohkuma T, Jun M, Rodgers A, Cooper ME, Glasziou P, Hamet P, Harrap S, Mancia G, Marre M, Neal B, Perkovic V, Poulter N, Williams B, Zoungas S, Chalmers J, Woodward M; ADVANCE Collaborative Group. Acute Increases in Serum Creatinine After Starting Angiotensin-Converting Enzyme Inhibitor-Based Therapy and Effects of its Continuation on Major Clinical Outcomes in Type 2 Diabetes Mellitus. Hypertension. 2019 Jan;73(1):84-91. doi: 10.1161/HYPERTENSIONAHA.118.12060. PMID 30571562
- [Derived] Thomas MC, Woodward M, Li Q, Pickering R, Tikellis C, Poulter N, Cooper ME, Marre M, Zoungas S, Chalmers J; ADVANCE Collaborative Group. Relationship Between Plasma 8-OH-Deoxyguanosine and Cardiovascular Disease and Survival in Type 2 Diabetes Mellitus: Results From the ADVANCE Trial. J Am Heart Assoc. 2018 Jun 30;7(13):e008226. doi: 10.1161/JAHA.117.008226. PMID 29960985
- [Derived] Welsh P, Rankin N, Li Q, Mark PB, Wurtz P, Ala-Korpela M, Marre M, Poulter N, Hamet P, Chalmers J, Woodward M, Sattar N. Circulating amino acids and the risk of macrovascular, microvascular and mortality outcomes in individuals with type 2 diabetes: results from the ADVANCE trial. Diabetologia. 2018 Jul;61(7):1581-1591. doi: 10.1007/s00125-018-4619-x. Epub 2018 May 4. PMID 29728717
- [Derived] Alshehry ZH, Mundra PA, Barlow CK, Mellett NA, Wong G, McConville MJ, Simes J, Tonkin AM, Sullivan DR, Barnes EH, Nestel PJ, Kingwell BA, Marre M, Neal B, Poulter NR, Rodgers A, Williams B, Zoungas S, Hillis GS, Chalmers J, Woodward M, Meikle PJ. Plasma Lipidomic Profiles Improve on Traditional Risk Factors for the Prediction of Cardiovascular Events in Type 2 Diabetes Mellitus. Circulation. 2016 Nov 22;134(21):1637-1650. doi: 10.1161/CIRCULATIONAHA.116.023233. Epub 2016 Oct 18. PMID 27756783
- [Derived] Mohammedi K, Woodward M, Zoungas S, Li Q, Harrap S, Patel A, Marre M, Chalmers J; ADVANCE Collaborative Group. Absence of Peripheral Pulses and Risk of Major Vascular Outcomes in Patients With Type 2 Diabetes. Diabetes Care. 2016 Dec;39(12):2270-2277. doi: 10.2337/dc16-1594. Epub 2016 Sep 27. PMID 27679583
- [Derived] van der Leeuw J, Visseren FL, Woodward M, van der Graaf Y, Grobbee DE, Harrap S, Heller S, Mancia G, Marre M, Poulter N, Zoungas S, Chalmers J. Estimation of individual beneficial and adverse effects of intensive glucose control for patients with type 2 diabetes. Diabetologia. 2016 Dec;59(12):2603-2612. doi: 10.1007/s00125-016-4082-5. Epub 2016 Sep 1. PMID 27586250
- [Derived] Mohammedi K, Woodward M, Hirakawa Y, Zoungas S, Williams B, Lisheng L, Rodgers A, Mancia G, Neal B, Harrap S, Marre M, Chalmers J; ADVANCE Collaborative Group. Microvascular and Macrovascular Disease and Risk for Major Peripheral Arterial Disease in Patients With Type 2 Diabetes. Diabetes Care. 2016 Oct;39(10):1796-803. doi: 10.2337/dc16-0588. Epub 2016 Jul 25. PMID 27456835
- [Derived] Hayes A, Arima H, Woodward M, Chalmers J, Poulter N, Hamet P, Clarke P. Changes in Quality of Life Associated with Complications of Diabetes: Results from the ADVANCE Study. Value Health. 2016 Jan;19(1):36-41. doi: 10.1016/j.jval.2015.10.010. Epub 2015 Dec 2. PMID 26797234
- [Derived] Blomster JI, Woodward M, Zoungas S, Hillis GS, Harrap S, Neal B, Poulter N, Mancia G, Chalmers J, Huxley R. The harms of smoking and benefits of smoking cessation in women compared with men with type 2 diabetes: an observational analysis of the ADVANCE (Action in Diabetes and Vascular Disease: Preterax and Diamicron modified release Controlled Evaluation) trial. BMJ Open. 2016 Jan 8;6(1):e009668. doi: 10.1136/bmjopen-2015-009668. PMID 26747037
- [Derived] Thomas MC, Woodward M, Neal B, Li Q, Pickering R, Marre M, Williams B, Perkovic V, Cooper ME, Zoungas S, Chalmers J, Hillis GS; ADVANCE Collaborative Group. Relationship between levels of advanced glycation end products and their soluble receptor and adverse outcomes in adults with type 2 diabetes. Diabetes Care. 2015 Oct;38(10):1891-7. doi: 10.2337/dc15-0925. Epub 2015 Aug 7. PMID 26253728
- [Derived] van der Leeuw J, Visseren FL, Woodward M, Zoungas S, Kengne AP, van der Graaf Y, Glasziou P, Hamet P, MacMahon S, Poulter N, Grobbee DE, Chalmers J. Predicting the effects of blood pressure-lowering treatment on major cardiovascular events for individual patients with type 2 diabetes mellitus: results from Action in Diabetes and Vascular Disease: Preterax and Diamicron MR Controlled Evaluation. Hypertension. 2015 Jan;65(1):115-21. doi: 10.1161/HYPERTENSIONAHA.114.04421. Epub 2014 Oct 13. PMID 25312436
- [Derived] Welsh P, Woodward M, Hillis GS, Li Q, Marre M, Williams B, Poulter N, Ryan L, Harrap S, Patel A, Chalmers J, Sattar N. Do cardiac biomarkers NT-proBNP and hsTnT predict microvascular events in patients with type 2 diabetes? Results from the ADVANCE trial. Diabetes Care. 2014 Aug;37(8):2202-10. doi: 10.2337/dc13-2625. Epub 2014 May 30. PMID 24879844
- [Derived] Hirakawa Y, Arima H, Zoungas S, Ninomiya T, Cooper M, Hamet P, Mancia G, Poulter N, Harrap S, Woodward M, Chalmers J. Impact of visit-to-visit glycemic variability on the risks of macrovascular and microvascular events and all-cause mortality in type 2 diabetes: the ADVANCE trial. Diabetes Care. 2014 Aug;37(8):2359-65. doi: 10.2337/dc14-0199. Epub 2014 May 8. PMID 24812434
- [Derived] Lowe G, Woodward M, Hillis G, Rumley A, Li Q, Harrap S, Marre M, Hamet P, Patel A, Poulter N, Chalmers J. Circulating inflammatory markers and the risk of vascular complications and mortality in people with type 2 diabetes and cardiovascular disease or risk factors: the ADVANCE study. Diabetes. 2014 Mar;63(3):1115-23. doi: 10.2337/db12-1625. Epub 2013 Nov 12. PMID 24222348
- [Derived] Hata J, Arima H, Rothwell PM, Woodward M, Zoungas S, Anderson C, Patel A, Neal B, Glasziou P, Hamet P, Mancia G, Poulter N, Williams B, Macmahon S, Chalmers J; ADVANCE Collaborative Group. Effects of visit-to-visit variability in systolic blood pressure on macrovascular and microvascular complications in patients with type 2 diabetes mellitus: the ADVANCE trial. Circulation. 2013 Sep 17;128(12):1325-34. doi: 10.1161/CIRCULATIONAHA.113.002717. Epub 2013 Aug 7. PMID 23926207
- [Derived] Blomster JI, Chow CK, Zoungas S, Woodward M, Patel A, Poulter NR, Marre M, Harrap S, Chalmers J, Hillis GS. The influence of physical activity on vascular complications and mortality in patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2013 Nov;15(11):1008-12. doi: 10.1111/dom.12122. Epub 2013 Jun 11. PMID 23675676
- [Derived] Zaman MJ, Patel A, Chalmers J, Woodward M, Clarke P, Li Q, Zoungas S. The effects of patient characteristics and geographical region on hospitalization in patients with type 2 diabetes. Diabet Med. 2013 Aug;30(8):918-25. doi: 10.1111/dme.12181. Epub 2013 Apr 12. PMID 23534416
- [Derived] Hata J, Arima H, Zoungas S, Fulcher G, Pollock C, Adams M, Watson J, Joshi R, Kengne AP, Ninomiya T, Anderson C, Woodward M, Patel A, Mancia G, Poulter N, MacMahon S, Chalmers J, Neal B; ADVANCE Collaborative Group. Effects of the endpoint adjudication process on the results of a randomised controlled trial: the ADVANCE trial. PLoS One. 2013;8(2):e55807. doi: 10.1371/journal.pone.0055807. Epub 2013 Feb 4. PMID 23390553
- [Derived] Hillis GS, Hata J, Woodward M, Perkovic V, Arima H, Chow CK, Zoungas S, Patel A, Poulter NR, Mancia G, Williams B, Chalmers J. Resting heart rate and the risk of microvascular complications in patients with type 2 diabetes mellitus. J Am Heart Assoc. 2012 Oct;1(5):e002832. doi: 10.1161/JAHA.112.002832. Epub 2012 Oct 25. PMID 23316296
- [Derived] Morton J, Zoungas S, Li Q, Patel AA, Chalmers J, Woodward M, Celermajer DS, Beulens JW, Stolk RP, Glasziou P, Ng MK; ADVANCE Collaborative Group. Low HDL cholesterol and the risk of diabetic nephropathy and retinopathy: results of the ADVANCE study. Diabetes Care. 2012 Nov;35(11):2201-6. doi: 10.2337/dc12-0306. Epub 2012 Aug 13. PMID 22891258
- [Derived] Wong G, Zoungas S, Lo S, Chalmers J, Cass A, Neal B, Woodward M, Perkovic V, Glasziou P, Williams B, Howard K, Chapman JR, Craig JC. The risk of cancer in people with diabetes and chronic kidney disease. Nephrol Dial Transplant. 2012 Aug;27(8):3337-44. doi: 10.1093/ndt/gfs022. Epub 2012 Feb 21. PMID 22357699
- [Derived] Zoungas S, Chalmers J, Ninomiya T, Li Q, Cooper ME, Colagiuri S, Fulcher G, de Galan BE, Harrap S, Hamet P, Heller S, MacMahon S, Marre M, Poulter N, Travert F, Patel A, Neal B, Woodward M; ADVANCE Collaborative Group. Association of HbA1c levels with vascular complications and death in patients with type 2 diabetes: evidence of glycaemic thresholds. Diabetologia. 2012 Mar;55(3):636-43. doi: 10.1007/s00125-011-2404-1. Epub 2011 Dec 21. PMID 22186981
- [Derived] Woodward M, Patel A, Zoungas S, Liu L, Pan C, Poulter N, Januszewicz A, Tandon N, Joshi P, Heller S, Neal B, Chalmers J. Does glycemic control offer similar benefits among patients with diabetes in different regions of the world? Results from the ADVANCE trial. Diabetes Care. 2011 Dec;34(12):2491-5. doi: 10.2337/dc11-0755. Epub 2011 Oct 4. PMID 21972410
- [Derived] Stefansdottir G, Zoungas S, Chalmers J, Kengne AP, Knol MJ, Leufkens HG, Patel A, Woodward M, Grobbee DE, De Bruin ML. Intensive glucose control and risk of cancer in patients with type 2 diabetes. Diabetologia. 2011 Jul;54(7):1608-14. doi: 10.1007/s00125-011-2104-x. Epub 2011 Apr 21. PMID 21509444
- [Derived] Zoungas S, Patel A, Chalmers J, de Galan BE, Li Q, Billot L, Woodward M, Ninomiya T, Neal B, MacMahon S, Grobbee DE, Kengne AP, Marre M, Heller S; ADVANCE Collaborative Group. Severe hypoglycemia and risks of vascular events and death. N Engl J Med. 2010 Oct 7;363(15):1410-8. doi: 10.1056/NEJMoa1003795. PMID 20925543
- [Derived] Glasziou PP, Clarke P, Alexander J, Rajmokan M, Beller E, Woodward M, Chalmers J, Poulter N, Patel A. Cost-effectiveness of lowering blood pressure with a fixed combination of perindopril and indapamide in type 2 diabetes mellitus: an ADVANCE trial-based analysis. Med J Aust. 2010 Sep 20;193(6):320-4. doi: 10.5694/j.1326-5377.2010.tb03941.x. PMID 20854235
- [Derived] Ninomiya T, Zoungas S, Neal B, Woodward M, Patel A, Perkovic V, Cass A, Cooper M, Grobbee D, Hamet P, Harrap S, Liu L, Mancia G, Mogensen CE, Poulter N, Rodgers A, Williams B, MacMahon S, Chalmers J; ADVANCE Collaborative Group. Efficacy and safety of routine blood pressure lowering in older patients with diabetes: results from the ADVANCE trial. J Hypertens. 2010 Jun;28(6):1141-9. PMID 20486273
- [Derived] Chalmers J, Arima H. Importance of blood pressure lowering in type 2 diabetes: focus on ADVANCE. J Cardiovasc Pharmacol. 2010 Apr;55(4):340-7. doi: 10.1097/fjc.0b013e3181d26469. PMID 20422738
- [Derived] Meier M, Hummel M. Cardiovascular disease and intensive glucose control in type 2 diabetes mellitus: moving practice toward evidence-based strategies. Vasc Health Risk Manag. 2009;5:859-71. doi: 10.2147/vhrm.s4808. Epub 2009 Nov 2. PMID 19898642
- [Derived] de Galan BE, Zoungas S, Chalmers J, Anderson C, Dufouil C, Pillai A, Cooper M, Grobbee DE, Hackett M, Hamet P, Heller SR, Lisheng L, MacMahon S, Mancia G, Neal B, Pan CY, Patel A, Poulter N, Travert F, Woodward M; ADVANCE Collaborative group. Cognitive function and risks of cardiovascular disease and hypoglycaemia in patients with type 2 diabetes: the Action in Diabetes and Vascular Disease: Preterax and Diamicron Modified Release Controlled Evaluation (ADVANCE) trial. Diabetologia. 2009 Nov;52(11):2328-2336. doi: 10.1007/s00125-009-1484-7. Epub 2009 Aug 18. PMID 19688336
- [Derived] Zoungas S, de Galan BE, Ninomiya T, Grobbee D, Hamet P, Heller S, MacMahon S, Marre M, Neal B, Patel A, Woodward M, Chalmers J; ADVANCE Collaborative Group; Cass A, Glasziou P, Harrap S, Lisheng L, Mancia G, Pillai A, Poulter N, Perkovic V, Travert F. Combined effects of routine blood pressure lowering and intensive glucose control on macrovascular and microvascular outcomes in patients with type 2 diabetes: New results from the ADVANCE trial. Diabetes Care. 2009 Nov;32(11):2068-74. doi: 10.2337/dc09-0959. Epub 2009 Aug 3. PMID 19651921
- [Derived] Beulens JW, Patel A, Vingerling JR, Cruickshank JK, Hughes AD, Stanton A, Lu J, McG Thom SA, Grobbee DE, Stolk RP; AdRem project team; ADVANCE management committee. Effects of blood pressure lowering and intensive glucose control on the incidence and progression of retinopathy in patients with type 2 diabetes mellitus: a randomised controlled trial. Diabetologia. 2009 Oct;52(10):2027-36. doi: 10.1007/s00125-009-1457-x. Epub 2009 Jul 25. PMID 19633827
- [Derived] de Galan BE, Perkovic V, Ninomiya T, Pillai A, Patel A, Cass A, Neal B, Poulter N, Harrap S, Mogensen CE, Cooper M, Marre M, Williams B, Hamet P, Mancia G, Woodward M, Glasziou P, Grobbee DE, MacMahon S, Chalmers J; ADVANCE Collaborative Group. Lowering blood pressure reduces renal events in type 2 diabetes. J Am Soc Nephrol. 2009 Apr;20(4):883-92. doi: 10.1681/ASN.2008070667. Epub 2009 Feb 18. PMID 19225038
- [Derived] ADVANCE Collaborative Group; Patel A, MacMahon S, Chalmers J, Neal B, Billot L, Woodward M, Marre M, Cooper M, Glasziou P, Grobbee D, Hamet P, Harrap S, Heller S, Liu L, Mancia G, Mogensen CE, Pan C, Poulter N, Rodgers A, Williams B, Bompoint S, de Galan BE, Joshi R, Travert F. Intensive blood glucose control and vascular outcomes in patients with type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2560-72. doi: 10.1056/NEJMoa0802987. Epub 2008 Jun 6. PMID 18539916
- [Derived] Patel A; ADVANCE Collaborative Group; MacMahon S, Chalmers J, Neal B, Woodward M, Billot L, Harrap S, Poulter N, Marre M, Cooper M, Glasziou P, Grobbee DE, Hamet P, Heller S, Liu LS, Mancia G, Mogensen CE, Pan CY, Rodgers A, Williams B. Effects of a fixed combination of perindopril and indapamide on macrovascular and microvascular outcomes in patients with type 2 diabetes mellitus (the ADVANCE trial): a randomised controlled trial. Lancet. 2007 Sep 8;370(9590):829-40. doi: 10.1016/S0140-6736(07)61303-8. PMID 17765963